CLINICAL TRIAL: NCT01425866
Title: Multicenter Randomized Trial of Structured Educational Intervention at the Community Level in Insufficiently Controlled Patients With Type 2 Diabetes in Reunion Island
Brief Title: Two Years Maintenance of Structured Group Self-management Education in Type 2 Diabetes : a Randomized Controlled Trial
Acronym: ERMIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010/CHR/03
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Structured self-management education; Therapeutic patient education; Lifestyle changes; Self-management Blood glucose; Empowerment; Adult learning; Socio-constructivism; Health management network; Reunion island
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 years self management education (Experimental): Long-term program including initial self-management education program (1 to 7 sessions, based on individual assessment), and follow-up group sessions maintained for 2 years (4-monthly assessment, empowerment, and contextual action planning; facultative additional specific thematic sessions being delivered if needed).
  Interventions: Behavioral: Structured self-management group education during 2 years
- Initial self-management education (Active Comparator): Initial self-management group education: 1 to 7 sessions (< 3 months), based on individual assessment.
  Interventions: Behavioral: Structured self-management group education during 2 years

INTERVENTIONS:
Behavioral: Structured self-management group education during 2 years — After an initial intensive group education, four-monthly follow-up self-management group education sessions for 2 years. Each session is based on empowerment, socio-constructivism, social learning theory: personalized assessment (BG and risk factors, actions: realized, planned, achieved (or not), cognitive work, analysis of individual and social context and environment (facilitators, obstacles) then action planning. Specific additional sessions can be scheduled (food management, diabetes treatment and hypoglycemia, exercise, self monitoring of BG, insulin dosage, foot care). Sessions are framed, and structured, with patient booklet support. Sessions are delivered at the community level, by trained registered nurses, under the coordination of the health management network Reucare.

SUMMARY:
Type 2 diabetes has a growing impact on populations and public health worldwide. Clinical trials have clearly demonstrated that a better control of blood glucose level and of other risk factors is efficient in preventing or retarding the complications of the disease. On Reunion island, Type 2 diabetes is present in 18% of population aged 30 or older with a high level of socio-economic deprivation. The hypothesis of the ERMIES study is that a structured group self-management education maintained at the community level for 2 years in patients with insufficiently controlled type 2 diabetes has better metabolic results (as attested by improvement in HbA1c level) at 2 yrs, compared to an initial short term (< 3 months) self-management program, based on the same theoretical basis and framework (learning nests empowerment). A total of 240 adults living in Reunion Island, with type 2 diabetes mellitus with HbA1c ≥ 7.5% on a stable treatment for at least 3 months will be randomly allocated to 2 intervention arms: either a short term (< 3 months) program (1 to 7 thematic 2-hr long sessions depending on individual assessment), or a long term program including the same initial program as 1st arm, but with group self management education sessions, maintained for 2 years (4-monthly assessment, empowerment, and contextual action planning; facultative additional specific thematic sessions being delivered if needed). Medical visits will be held quarterly for the recording of outcome measures (HbA1c, blood pressure, anthropometrics, tobacco consumption, diabetes complications) and yearly for blood glucose, lipids, micro-albuminuria or proteinuria, creatinine clearance, diet and exercise (questionnaires), treatment recording, quality of life, self-efficacy, anxiety and depression scales, and social support.

DETAILED DESCRIPTION:
Randomised clinical trial comparing 2 parallel arms of educational intervention with the hypothesis of the superiority of a 2-year maintenance of a structured, theoretically-based, educational follow-up. All subjects of both arms will beneficiate from an initial structured educational program (< 3-months). Subjects, educators, and investigators will be unaware of the group allocation during this initial round. Then the intervention arm will undergo a 2 years self management educational follow-up program. Randomisation will be stratified on 2 factors : centres (5 strata) and anti diabetic treatment (2 strata: insulin-treated or not). All group sessions (3-10 subjects, 2 hr-long, one assessment group session and 6 facultative additional specific sessions for each round [initial in both arms or follow-up in the intervention arm], as needed and planned during the first) will be held at the community level, as closer as possible to the subjects' residence. Educators are specifically trained and the educational sessions are structured and coordinated in the framing and organisational supervision of the health management network "ReuCARE" in Reunion island. Subjects of both arms will continue quarterly to attend at the outpatient clinic of the centre. This trial is associated to a qualitative ethno-sociological study on a sample of 30-40 subjects, with in-depth interviews and ethnographic observation of group sessions, with the specific aim of describing the learning processes, coping, health and functional literacy, social and contextual issues.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c ≥ 7,5% more than 3 months
* Adults
* ≥ 1 year ADO and/or insulin and/or GLP-1 analog
* antidiabetic treatment unchanged since 3 months (no change of treatment in the last 3 months, except for insulin dosage)
* Living in Reunion Island
* Affiliated to French national health insurance
* Signed informed consent

Exclusion Criteria:

* Treatment or associated conditions that would influence glycemic control, such as corticotherapy, cancer, inflammatory chronic diseases
* Hospitalisation linked to diabetes < 3 months
* Structured patient education in the past 3 months
* Severe diabetes complications (e.g. ischemic or proliferative retinopathy, severe renal failure (clearance < 15 ml/min), acute ischemic heart disease (< 6 months, foot lesion)
* Pregnancy (on-going or planned during the study)
* Evolutive cancer
* Physical or cognitive heavy handicap
* Concomitant participation to a therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mean change in glycated haemoglobin (GlyHb) | 0 and 2 years

SECONDARY OUTCOMES:
Mean change in glycated haemoglobin (GlyHb) | 0 and 1 year
change in GlyHb | quarterly up to 2 yrs
Blood sugar and lipids | 1 and 2 yrs
  Blood sugar Total, HDL and LDL cholesterol, triglycerides
diabetes complications | 1 and 2 yrs
  retinopathy stages, micro-albuminuria or proteinuria, creatinine clearance, foot risk grade, ischemic heart or cerebral disease
health behaviours | 1 and 2 yrs
  physical activity and diet (Baecke and food frequency questionnaires)
anti-diabetic therapy | 1 and 2 yrs
  type, dosage
health care process | 1 and 2 yrs
  medical follow-up and appointments, compliance (questionnaire)
Psychometric scales | 1 and 2 yrs
  self-efficacy, social support, HAD (anxiety and depression)
Quality of Life | 1 and 2 yrs
  short DQOL adapted and validated for Reunion
Change in tobacco consumption | quarterly up to 2 yrs
Change in fasting blood glucose | quarterly up to 2 yrs
Change in body mass index | quarterly up to 2 yrs
Change in waist circumference | quarterly up to 2 yrs
Change in blood pressure | quarterly up to 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Debussche, MD, Principal Investigator — Diabetology - University Hospital Reunion Island - Felix Guyon Site; Jean Luc YVIN, MD, Principal Investigator — Department of Internal Medicine - University Hospital Reunion Island - Felix Guyon Site; Stéphane SCHNEEBELI, MD, Principal Investigator — Diabetology - University Hospital Reunion Island - GHSR; Jean Hugues GATINA, MD, Principal Investigator — Centre Hospitalier Gabriel Martin; Yogananda THIRAPATHIAPPADU, MD, Principal Investigator — Groupe Hospitalier Est Réunion
Locations (4):
- France (4):
  - Groupe Hopitalier Est Réunion, Saint-Benoît, La Réunion
  - Centre Hospitalier Gabriel Martin, Saint-Paul, La Réunion
  - Diabetolgy - UNiversity Hospital Sud Réunion, Saint-Pierre, La Réunion
  - Department of endocrinology, University Hospital Reunion Island - Felix Guyon Site, Saint Denis de La Réunion

REFERENCES:
- [Derived] Flaus-Furmaniuk A, Fianu A, Lenclume V, Chirpaz E, Balcou-Debussche M, Debussche X, Marimoutou C. Attrition and social vulnerability during 2-year-long structured care in type 2 diabetes, the ERMIES randomized controlled trial. BMC Endocr Disord. 2022 Dec 13;22(1):314. doi: 10.1186/s12902-022-01211-3. PMID 36510180
- [Derived] Debussche X, Balcou-Debussche M, Ballet D, Caroupin-Soupoutevin J. Health literacy in context: struggling to self-manage diabetes - a longitudinal qualitative study. BMJ Open. 2022 Jun 14;12(6):e046759. doi: 10.1136/bmjopen-2020-046759. PMID 35701054
- [Derived] Debussche X, Collin F, Fianu A, Balcou-Debussche M, Fouet-Rosiers I, Koleck M, Favier F. Structured self-management education maintained over two years in insufficiently controlled type 2 diabetes patients: the ERMIES randomised trial in Reunion Island. Cardiovasc Diabetol. 2012 Aug 2;11:91. doi: 10.1186/1475-2840-11-91. PMID 22856504